CLINICAL TRIAL: NCT06090097
Title: Knee-Biofeedback Rehabilitation Interface for Game-based Home Therapy
Brief Title: Knee Biofeedback Rehabilitation Through Game Therapy
Acronym: KneeBRIGHT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KneeBRIGHT2B
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis, physical therapy, rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Outcomes Assessor
Masking Description: Researchers conducting functional outcomes on study completion will be blinded from the intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- KneeBRIGHT Group (Experimental): The interventional group will conduct all exercises during the 10-week therapy regimen using the KneeBRIGHT electromyogram sensors and game software.
  Interventions: Device: KneeBRIGHT System
- Control Group (Active Comparator): The control group will conduct all exercises following a standard physical therapy regimen.
  Interventions: Other: Control Exercise

INTERVENTIONS:
Device: KneeBRIGHT System — The KneeBRIGHT system includes electromyogram sensors and video game software that leads participants through physical therapy exercise.
  Arms: KneeBRIGHT Group
Other: Control Exercise — The control group will complete a 10-week regimen of conventional PT exercise
  Arms: Control Group

SUMMARY:
The goal of this study is to learn about the effect of video-game based rehabilitation exercise for patients with knee osteoarthritis. The main question the study aims to answer is: do patients who exercise with the game have better functional outcomes and engagement compared to patients who do conventional exercise? Participants will complete 10 weeks of physical therapy exercise sessions that focus on quadriceps strengthening. Two sessions per week will be conducted in the clinic, and one session will be conducted at home each week. The interventional group will conduct all exercises using the KneeBRIGHT EMG sensors and game software. The control group will conduct all exercises following a standard physical therapy regimen. Researchers will compare knee function and engagement between the group who uses the game, and the group who does conventional exercise.

DETAILED DESCRIPTION:
The KneeBRIGHT game system will be evaluated in a 10-week single-blinded randomized controlled trial. The goals of this study are to: (1) assess improvements in functional outcomes following an exercise regimen conducted by KneeBRIGHT compared to conventional exercise; and (2) evaluate patient engagement during unsupervised, home-based exercises with and without the KneeBRIGHT software. Over the course of the study period, the knee OA participants will conduct physical therapy sessions with the physical therapist (PT) who enrolled them. The exercise regimen will implement each PT's standard of care, consisting of two weekly clinic sessions and one weekly home exercise session, for 10 weeks. Knee OA participants will be randomly assigned (via block randomization for each PT) to use either the KneeBRIGHT system for both clinic and home exercise, or to receive standard care with conventional exercise routines. Participants will conduct functional exercise assessments on study intake and again on study completion. Participants will also complete questionnaires focused on exercise engagement on study completion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis via x-ray, with a score of at least 2 (out of 4) on the Kellgren-Lawrence OA scoring system; independent ambulation without assistive device

Exclusion Criteria:

* individuals who have psychiatric or cognitive impairment (e.g., dementia) that interferes with their ability to follow instructions or provide voluntary consent; symptomatic spine, hip, ankle, or foot disease other than OA that would interfere with assessment of the knee.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score | After 10 weeks (study completion)
  A multi-dimensional assessment that classifies knee outcomes into five categories: pain, symptoms, activities of daily living (ADL), sport, and quality of life
Timed get-up-and-go score | After 10 weeks (study completion)
  In the timed up and go (TUG) test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again.
6-minute walk test | After 10 weeks (study completion)
  The six-minute walk test (6MWT) measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface.
Quadriceps strength | After 10 weeks (study completion)
  Quadriceps strength will be measured by recording isokinetic knee extension torque as measured by a dynamometer
Patient Activation Model Scores | After 10 weeks (study completion)
  The Patient Activation Model (PAM) is an established, highly reliable, questionnaire that reflects a developmental model of patient engagement with their healthcare regimens

SECONDARY OUTCOMES:
Patient technology acceptance | After 10 weeks (study completion)
  Participants will complete a questionnaire, designed based on the established Technology Acceptance Model to assess their level of technology acceptance.

OTHER OUTCOMES:
Patient home exercise adherence | After 10 weeks (study completion)
  The KneeBRIGHT software will log the exercises completed at home; these logs will report number of exercises conducted, level of resistance, and timestamps for the sessions. Control group participants will log home exercises using a written checklist of exercises

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Krepkovich, MS, Principal Investigator — Barron Associates
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No